CLINICAL TRIAL: NCT03572868
Title: Perinatal and Long-term Outcome of Newborns With an Isolated Small Transverse Cerebellar Diameter
Brief Title: Long-term Outcome of Newborns With an Isolated Small Cerebellum
Acronym: PECERI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0273
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Cerebellar Hypoplasia
MeSH Terms: conditions — Cerebellar Hypoplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of the long term neurodevelopmental outcome — Evaluation of the long-term neurodevelopmental outcome of newborns who have an isolated transverse cerebellar diameter < 5th centile during the second or the third trimester of pregnancy.

SUMMARY:
The decreased cerebellar biometry during second and third trimester ultrasound examination is the main parameter to diagnoses cerebellar and pontocerebellar hypoplasia. Investigators already described that a transverse cerebellar diameter (TCD) below the 5th centile at second or third trimester scan is related to a high rate of fetal malformations, severe intrauterine restriction in growth, chromosomal anomalies and genetic disorders, therefore when facing a TCD below the 5th centile, patients should be referred for oriented sonogram, fetal MRI (Magnetic resonance imaging) and fetal karyotyping.

However, prenatal counseling in case of an isolated decreased cerebellar biometry remains challenging since there are no data in the literature regarding the neurodevelopmental outcome of these newborns. The aim of this work is to evaluate the neurodevelopmental outcome of newborns with a prenatal isolated decreased cerebellar biometry, in order to improve prenatal counseling.

ELIGIBILITY:
Inclusion Criteria:

* 2nd or the 3rd trimester ultrasound examination realized at the hospital "Femme Mère Enfant" in Lyon between 2008 and 2015
* Isolated Transverse cerebellar diameter <5th centile
* Parents who received the information and did not object to participate to the study

Exclusion Criteria:

* Decreased Transverse cerebellar diameter with associated malformations diagnosed during prenatal period
* Family history of neurodevelopmental delay or cognitive impairment
* Preterm delivery (< 28 WG)
* Severe restriction in growth at birth (<3e centile)
* Neonatal asphyxia (pH blood cord < 7)
* Apgar score < 7 at 5 min of live with transfer to the neonatal intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of newborns who have an isolated transverse cerebellar diameter < 5th centile during the 2nd or the 3rd trimester ultrasound examination realized at the hospital Femme Mère Enfant in Lyon between 2008 and 2015.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Development Quotient. | between 3 and 10 years after birth
  Development Quotient of each child established from CDI questionnaire (Child Development Inventory).

CONTACTS AND LOCATIONS:
Locations (1):
- Service Obstétrique - Hôpital Femme Mère Enfant - Groupement Hospitalier Est, Bron, France

IPD SHARING:
Plan to Share IPD: No